CLINICAL TRIAL: NCT06505057
Title: Ovarian Tissue Cryopreservation and Subsequent Auto-Transplantation for Female
Brief Title: Ovarian Tissue Cryopreservation and Subsequent Auto-Transplantation for Female Cancer Patients (HKCH)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PAED-2023-079
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ovarian tissue freezing and subsequent auto-transplantation after thawing (Experimental): Removal of the ovarian tissue will be retrieved via laparoscopic surgery under general anesthesia. The ovarian cortical tissue obtained will be transferred on ice to the laboratory for cryopreservation. After medical treatment, if the patient would like to start a family but has experienced premature ovarian failure, she will have ovarian tissue auto-transplantation after thawing.
  Interventions: Other: Ovarian Tissue Cryopreservation and Subsequent Auto-Transplantation

INTERVENTIONS:
Other: Ovarian Tissue Cryopreservation and Subsequent Auto-Transplantation — Ovarian Tissue Cryopreservation and Subsequent Auto-Transplantation

SUMMARY:
Ovarian tissue freezing is an ideal option for these patients as it can be performed immediately and does not need any time for ovarian stimulation. We hope we can develop this service in our locality to allow more young female cancer patients to have their fertility preserved.

DETAILED DESCRIPTION:
To date, transplantation of cryopreserved ovarian tissue has resulted in births of at least 130 children but data on transplantation of ovarian tissue removed before puberty are scarce.

During ovarian tissue cryopreservation (OTC), it is possible to freeze isolated oocytes. In 2003, Revel et al described for the first time oocyte isolation in children younger than 12 years with seven, eight and seven oocytes isolated from the ovarian cortex of patients aged 5, 8 and 10 years, respectively.

At this moment, financial constraint is another great hindrance to fertility preservation in Hong Kong as the procedure is not cheap. Cryopreservation of gametes and embryos involving assisted reproductive technology is expensive and the costs of fertility preservation impose a great burden to these cancer patients on top of the great expenses for their chemo- or radiotherapy. It is almost impossible for underprivileged families.

Young cancer patients may often need immediate gonadotoxic treatment for their cancer, just like those with haematological cancers. In these patients, egg or embryo freezing is not possible as it takes at least 8-12 days' time for ovarian stimulation. Ovarian tissue freezing is an ideal option for these patients as it can be performed immediately and does not need any time for ovarian stimulation. We hope we can develop this service in our locality to allow more young female cancer patients to have their fertility preserved.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 0-35 years old and diagnosed with cancer e.g., leukaemia, myeloproliferative or myelodysplastic diseases, lymphoma, bone tumours, neurological neoplasms and sarcoma, Paediatric bone marrow transplant patients
* Patients with any illness or who will undergo any type of treatment that may cause irreversible damage to their fertility, such as extensive abdominal surgery, high toxicity medication and treatments;
* Patients suffering from hormone-sensitive malignancies who will undergo medical treatment, such as radiotherapy and chemotherapy that is liable to damage their ovaries and deter them from conception in the future.

Exclusion Criteria:

Patients with no anticipated oncologic therapies Patients who are pregnant Children with one ovary Children deemed high risk for perioperative complications Patients unable to provide consent/assent (i.e. significant psychiatric problems/cognitive delay)

-

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2039-07-31 (Estimated); Study Completion 2041-07-31 (Estimated)

PRIMARY OUTCOMES:
Surgical complications | 15 years
  Surgical complications after ovarian tissue transplantation

SECONDARY OUTCOMES:
Pregnancy rate | 15 years
  Pregnancy rate after ovarian tissue transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Pui Wah CHUNG, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No